CLINICAL TRIAL: NCT01206010
Title: Effects of a Tailored Dose of Varenicline on Post-quitting Urges to Smoke
Brief Title: Tailoring Varenicline to Individual Needs (TVIN Study)
Acronym: TVIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Dr. Al-Rehan Abdul Aziz Dhanji, Clinical Fellow in Cardiothoracic Surgery, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: qmul010610; 2010-022335-11 (EudraCT Number)
Record Dates: First submitted 2010-09-14; First posted 2010-09-21 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Tobacco Dependence; Smoking Cessation
Keywords: Tobacco Dependence; Smoking cessation; Varenicline; Tailored dosing
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline + Active Tailored Dose (Experimental)
  Interventions: Drug: Varenicline
- Varenicline + Placebo Tailored Dose (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Participants will increase varenicline dose by 0.5 mg twice daily every three days to a maximum of 2.5 mg twice daily. This increased dose will be continued for 3-weeks before being reduced to the standard dose of 1.0 mg twice daily.
  Other Names: Champix; Chantix
  Arms: Varenicline + Active Tailored Dose
Drug: Placebo — Participants will increase placebo dose by 0.5 mg twice daily every three days to a maximum of 2.5 mg twice daily. This increased dose will be continued for 3-weeks before being reduced to the standard varenicline dose of 1.0 mg twice daily.
  Other Names: Champix; Chantix
  Arms: Varenicline + Placebo Tailored Dose
Drug: Varenicline — All participants will receive the standard dose of Varenicline (14 weeks): 0.5 mg once daily for days 1-3, 0.5 mg twice daily for days 4-7, and then a continuation dose of 1.0 mg twice daily. In addition to this participants will use an tailored varenicline/placebo dose up to maximum of 2.5 mg twice daily for 3 weeks.
  Other Names: Champix; Chantix

SUMMARY:
Varenicline is a partial nicotinic agonist which acts on alpha4 beta2 nicotinic receptors. It is presumed to alleviate withdrawal discomfort, but also to diminish rewarding effects of cigarettes. The standard varenicline dosing has been formulated to avoid adverse reactions (primarily nausea) in sensitive clients. The downside of this cautious approach is that a substantial proportion of clients may be under-dosed. A blanket dose increase would inevitably increase the incidence of side effects, but it is likely that tailoring varenicline dosing to clients' needs would be safe and may further increase varenicline's efficacy.

This study will recruit 200 smokers who report little change to their enjoyment of cigarettes and no nausea, during the first week of varenicline use. These smokers will be randomised to receive the standard dose plus placebo or plus individualised varenicline dose up to 5mg, titrated over the next week prior to their target quit day. Urges to smoke, and other withdrawal symptoms, experienced during the study period will be compared between groups to see if the tailored therapy may be useful.

ELIGIBILITY:
Inclusion Criteria:

* Smoker seeking treatment
* Aged 18 and over
* Consenting to take part
* Report little or no change in enjoyment of cigarettes and/or nausea

Exclusion Criteria:

* Pregnant or breastfeeding
* Have severe kidney disease
* Have severe heart problems
* Have a current psychiatric illness
* Are unable to fill in questionnaires in English
* Have an allergy to varenicline
* Are currently involved in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Rating of urges to smoke 1-week after the target quit | 1 week
  Rating of urges to smoke will be assessed using the Mood & Physical Symptoms Scale

SECONDARY OUTCOMES:
Identification of the number of people with no effect of varenicline (as measured on a self reported questionnaire) prior to the target quit date | 2 weeks pre quitting
The change of withdrawal symptoms from target quit day over the first 4-weeks of abstinence assessed by the Mood and Physical Symptoms Scale | 4 weeks post quitting
Validated abstinence rates at 1-12 weeks post target quit date | 1-12 weeks post target quit date
Profile of all adverse effects (as measured by a self reported questionnaire) reported up to 12-weeks post quitting | Up to 12 weeks post quitting
Client ratings (measured using a self-reporting questionnaire) of tailored treatment regimen | Up to 12 weeks post quit
Rating of urges to smoke 24 hours post target quit date | 24 hours post target quit date

CONTACTS AND LOCATIONS:
Overall Officials: Al-Rehan Abdul Aziz Dhanji, MB.BS., BSc.,MRCS., Principal Investigator — Queen Mary University of London
Locations (1):
- Tobacco Dependence Research and Treatment Unit, London, United Kingdom

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hajek P, McRobbie H, Myers Smith K, Phillips A, Cornwall D, Dhanji AR. Increasing varenicline dose in smokers who do not respond to the standard dosage: a randomized clinical trial. JAMA Intern Med. 2015 Feb;175(2):266-71. doi: 10.1001/jamainternmed.2014.6916. PMID 25545858